CLINICAL TRIAL: NCT01600287
Title: Evaluation of Closed Loop Anaesthesia Delivery System for Propofol Anaesthesia in Pediatric Cardiac Surgery
Brief Title: Closed Loop Propofol Administration in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, INDRANIL BISWAS, Indranil Biswas, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 8450/PG-2Trg/2010/
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-07

CONDITIONS: Pediatric Cardiac Surgery; Intraoperative Awareness; Automated Drug Delivery
Keywords: bispectral index; propofol; paediatric cardiac surgery; closed loop anaesthesia delivery system
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAADS group (Experimental): dosage of propofol adjusted automatically by IAADS
  Interventions: Other: IAADS
- Manual group (Active Comparator): dosage of propofol adjusted manually
  Interventions: Other: Manual propofol administration

INTERVENTIONS:
Other: IAADS — In automatic mode, the system requests an update of the BIS data every 5 seconds and calculates the BIS "error" (difference between the target and actual BIS value). This value along with the trends of BIS in the epoch of the last 30 seconds as well as in the last 5 minutes is passed on to a patient individualized, model based adaptive control algorithm. The algorithm uses the error to calculate an adjustment to the propofol delivery rate, but does not apply it immediately. Adjustments to the propofol delivery rate are only made every 30 seconds, taking into account the sum of previous six BIS "error" values, the trends of BIS in the epoch of last 30 seconds as well as in the last 5 minutes, time elapsed since the initiation of infusion, pharmacokinetics, the time delay factor between sensing and averaging of BIS data, the time delay factor between the change in infusion rate and the actual change in the plasma concentration of propofol as well as the peak effect of propofol.
  Arms: IAADS group
Other: Manual propofol administration — In "manual" mode, the user can also control the propofol infusion rate manually, using the keyboard or the mouse of the PC. The PC displays a graph of the propofol delivery rate and trend of BIS value.
  Arms: Manual group

SUMMARY:
The purpose of the study is to evaluate and compare the feasibility, efficacy and safety of IAADS (Improved Anaesthetic Agent Delivery System) for propofol anaesthesia against manual control using bispectral index in paediatric patients undergoing open heart surgery under cardio-pulmonary bypass.

DETAILED DESCRIPTION:
Automated drug delivery has gained considerable interest in recent times. It is carried out by specially programmed electro-mechanical devices where dose rate adjustment is made independent of human intervention. The desired target is chosen by the clinician. The closed loop system depends upon a feedback signal to modify the rate of drug delivery. These have an advantage that they are able to overcome the individual pharmacokinetic and pharmacodynamic differences as well as the differing levels of surgical stimulation. Majority of studies on closed loop delivery of hypnotics has been done using propofol. CLADS(Closed loop anesthesia delivery system) is a BIS guided closed loop anaesthesia delivery system developed at PGIMER (Post graduate institute of medical education and research), Chandigarh and has been used successfully for administration of propofol in various situations, eg, non-cardiac surgery, cardiac surgery, post-operative sedation and high altitude. The system used will be IAADS, Improved anesthetic agent delivery system - the present and updated version of CLADS), a pharmacokinetic-pharmacodynamic model based adaptive system . There are only a few studies/reports regarding closed loop delivery of muscle relaxants in children. In this study, the efficacy of IAADS will be compared with manual control for administration of propofol using BIS as a control variable during induction and maintenance of anaesthesia in children undergoing elective open heart surgery.

After approval from the Institutional ethics committee and written informed parental consent, 40 children, aged 5-18 years and ASA physical status II-III, planned for elective open heart surgery under general anaesthesia will be studied. Patients will be randomly allocated to one of two groups - the manual group and the IAADS group using computer-generated random numbers in sealed opaque envelopes. Exclusion criteria will be: patients weighing more than ±30% of ideal body weight, those with neurological/psychological disorders, on psychoactive medications, belonging to NYHA class IV, those with severe stenotic valvular lesions, with known allergy to propofol or any of its constituents, having severe pulmonary arterial hypertension, with cyanotic congenital heart disease and those who may require deep hypothermic circulatory arrest for repair. The investigator will be present during the procedure for data collection purpose only and was not involved in the conduct of anaesthesia. Patients will be premedicated with oral midazolam syrup 0.25mg/kg 30 minutes before shifting to operating room. EMLA cream will be applied to the site of venipuncture for at least one hour. Intravenous access will be obtained in the operating room. Routine physiological monitoring will be commenced (pulse oximetry, electrocardiography, non-invasive blood pressure). BIS will be obtained by disposable sensors (Aspect Medical System Inc. MA USA) attached to the forehead of the patients. The children resisting venous cannula placement will be excluded from the study and subjected to inhalational induction.

Before induction, patients will receive fentanyl 3µg/kg over three minutes. In automatic mode, IAADS will calculate and titrate the initial and subsequent propofol infusion rate according to the weight of the patient, the risk status, the target BIS value which will be set at 50 for all cases. In manual mode, infusion rate will be determined by the attending anaesthesiologist according to the weight of the patient and target BIS of 50, with the aim to maintain BIS within 40-60. After loss of consciousness, patients will receive 0.1mg/kg of vecuronium bromide and trachea will be intubated after 4 minutes. The lungs will be ventilated with 100% O2; tidal volume and respiratory rate will be adjusted to maintain an EtCO2 of 30-35 mm Hg. Central venous catheter and arterial cannula will be inserted subsequently.

Analgesia will be maintained with infusion of fentanyl at 1µg/kg/hr and additional boluses of 1µg/kg will be administered before skin incision, sternotomy and commencement of cardio-pulmonary bypass. Muscle relaxation will be maintained with vecuronium bromide. Tachycardia and hypertension will be treated with fentanyl bolus, esmolol, nitroglycerine as appropriate. Hypotension will be treated with fluid bolus, phenylephrine, inotropes as appropriate. Significant bradycardia will be treated with atropine sulphate. During CPB, infusion of fentanyl and propofol will be continued. MAP will be maintained between 30-50 mm Hg and any deviation from these limits will be treated with phenylephrine boluses or nitroglycerine infusion. Propofol will be administered as per IAADS protocol in automatic group and manually in control group. The number of times propofol infusion rate that will needed to be changed in the manual group will be noted.

After skin closure, fentanyl and propofol infusion will be stopped, study protocol will be terminated and the patients will be shifted to ICU without antagonizing the muscle relaxant for elective mechanical ventilation. Patients will be given propofol infusion for postoperative sedation and will be extubated when standard criteria for weaning and extubation will be met. The children will be subjected to a structured interview as described by Lopez et a for conscious awareness; on second day after surgery and approximately one month later.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 5-18 years and ASA (American Society of Anesthesiology) physical status 2-3, planned for elective open heart surgery under general anaesthesia.

Exclusion Criteria:

* Patients weighing more than ±30% of ideal body weight.
* Patients having neurological/psychological disorders or on psychoactive medications.
* Patients belonging to NYHA (New York Heart Association) class IV.
* Patients with severe stenotic valvular lesions, eg, mitral or aortic stenosis.
* Patients with known allergy to propofol or any of its constituents.
* Patients having severe pulmonary arterial hypertension.
* Patients with cyanotic congenital heart disease.
* Patients requiring deep hypothermic circulatory arrest during surgery.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indranil Biswas, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Goverdhan D Puri, MBBS,MD,PhD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Preethy J Mathew, MBBS,MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Advanced Cardiac Centre.Postgraduate Institute of Medical Education and Research., Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Agarwal J, Puri GD, Mathew PJ. Comparison of closed loop vs. manual administration of propofol using the Bispectral index in cardiac surgery. Acta Anaesthesiol Scand. 2009 Mar;53(3):390-7. doi: 10.1111/j.1399-6576.2008.01884.x. PMID 19243324
- [Background] Solanki A, Puri GD, Mathew PJ. Bispectral index-controlled postoperative sedation in cardiac surgery patients: a comparative trial between closed loop and manual administration of propofol. Eur J Anaesthesiol. 2010 Aug;27(8):708-13. doi: 10.1097/EJA.0b013e328335b2d4. PMID 20299990
- [Background] Puri GD, Kumar B, Aveek J. Closed-loop anaesthesia delivery system (CLADS) using bispectral index: a performance assessment study. Anaesth Intensive Care. 2007 Jun;35(3):357-62. doi: 10.1177/0310057X0703500306. PMID 17591128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 patients assessed in surgical ward between january 2012 to september 2012, after excluding 11 patients, 40 remaining patients were randomised into two groups(IAADS & Manual) of 20 each- all patients in each group received allocated interventions- no patients needed to be excluded from final analysis.
Pre-assignment Details: 5 patients were initially excluded because of having cyanotic heart disease, 6 patients excluded subsequently as they resisted pre-induction venous cannula placement.
Groups:
- IAADS Group: Both induction and maintenance of anesthesia was done automatically by IAADS according to age, sex, height of the patient, target BIS(50) entered, risk status and maximum allowable rate entered.
- Manual Group: dosage of propofol was adjusted manually by the attending anesthesiologist through the keyboard of the PC attached to the syringe pump for both induction and maintenance.
Period: Overall Study
Arm/Group | IAADS Group | Manual Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IAADS Group | Manual Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.1 (5.1) | 12 (4.1) | 11.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  India | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Bispectral Index(BIS) Remains+/-10 of Target
Description: The primary outcome to be measured is the ability of the system to keep the depth of anesthesia in the target range, i.e, Bispectral Index(BIS) value of 50+/- 10. This will assess the ability of the system to prevent intra-operative awareness of the patients and at the same time avoid excessive depth of anesthesia with its accompanying adverse effects.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
percentage of time | 77.4 (13.07) | 75 (11)

2. Secondary Outcome: Median Performance Error(MDPE)
Description: The difference between the observed and target of measure of depth of anesthesia (BIS) expressed as percentage of target BIS is calculated as performance error every 30 seconds. This value may be either '+' or '_' indicating whether the observed measure is above the target (overshoot-+) or below the target (undershoot-_). The median value of all performance errors during propofol anesthesia is median performance error and is a measure of bias of the system. This outcome is expressed as the mean of Median Performance Errors per participant.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: errors per participant
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
errors per participant | 6 (8) | -7 (5)

3. Secondary Outcome: Median Absolute Performance Error(MDAPE)
Description: The difference between the observed and target of measure of depth of anesthesia (BIS) expressed as percentage of target BIS is calculated as performance error every 30 seconds. This value may be either '+' or '_' indicating whether the observed measure is above the target (overshoot-+) or below the target (undershoot-_).The median of the absolute values of performance errors (without considering the direction of error) is median absolute performance error. This outcome measures the magnitude of error or inaccuracy of the system studied. A lower value indicates a more precise system.This outcome is expressed as the mean of Median Absolute Performance Errors per participant.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: errors per participant
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
errors per participant | 12 (3) | 13 (4)

4. Secondary Outcome: Wobble
Description: Wobble measures the intra-individual variability in performance error.The median of the difference between individual performance errors throughout anesthesia and the median performance error for each participant is the wobble of that participant. The mean value per participant is indicated in the outcome measure.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: errors per participant
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
errors per participant | 9 (3) | 11 (4)

5. Secondary Outcome: Percentage of Time Heart Rate Remains Within 25% of Pre-op Baseline
Description: The duration of time heart rate remains within 25% of the pre-operative baseline value during the period propofol (general anesthetic) is administered to the study population. This value is expressed as a percentage. This outcome is expressed as the mean of percentage of time per participant.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
percentage of time | 83.3 (11.7) | 80.5 (19.6)

6. Secondary Outcome: Percentage of Time Mean Arterial Pressure Remains Within 25% of Pre-op Baseline
Description: The duration of time mean arterial pressure remains within 25% of the pre-operative baseline value during the period propofol (general anesthetic) is administered to the study population. This value is expressed as percentage. This outcome is expressed as the mean of percentage of time per participant
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
percentage of time | 83.8 (10.5) | 72.8 (18.4)

7. Secondary Outcome: Intra-operative Awareness
Description: The number of patients who will be able to recall the intra-operative events when assessed postoperatively. This will be assessed by a structured protocol
Time Frame: Approximately 3 days and then 1 month later
Measure: Number; unit: participants
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

8. Secondary Outcome: Divergence
Description: slope of the linear regression curve of performance error against time.
Time Frame: 8 hours (approx)
Measure: Mean (Standard Deviation); unit: errors per second
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
errors per second | 0.02 (0.17) | -0.097 (0.219)

9. Secondary Outcome: Global Score
Description: overall performance assessment of the system calculated as= [(MDAPE+Wobble)/percentage of time BIS remains within target]x100 Lower score indicates better overall performance
Time Frame: 8 hours (approx)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
percentage of time | 30.09 (12.17) | 34.12 (15.28)

10. Secondary Outcome: Intraoperative Phenylephrine Used (Pre CPB)
Description: total phenylephrine dose needed to be used in the pre CPB period to maintain hemodynamic stability
Time Frame: 2 hours(approx)
Measure: Mean (Standard Deviation); unit: microgram per Kg body weight
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
microgram per Kg body weight | 5.79 (5.98) | 16.92 (10.92)

11. Other Pre Specified Outcome: Induction Dose of Propofol
Description: Dose of propofol needed for induction
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: mg per kg body weight
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
mg per kg body weight | 2.06 (0.79) | 2.95 (1.03)

12. Other Pre Specified Outcome: Induction Time
Description: Time required for the first time achievement of two subsequent BIS values below or equal to 55
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
seconds | 186.2 (91.2) | 160.6 (42)

13. Other Pre Specified Outcome: Minimum BIS During Induction
Description: Bispectral Index(BIS) is an EEG-based objective measure of anesthetic depth with values ranging from 100 to 0, lower number indicating greater depth of anesthesia. Values between 40 to 60 indicate adequate depth required for surgery. During induction of anesthesia, there is a tendency of overshooting the adequate depth of anesthesia, due to use of higher dose and rate of administration required for induction. The minimum BIS achieved during induction is a measure of this overshoot. The less the minimum value, the more is the overshoot, worse the outcome is. The minimum BIS during induction is automatically stored in the PC used for the study.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: Bispectral Index
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
Bispectral Index | 45 (6) | 36 (11)

14. Other Pre Specified Outcome: Percentage Fall in MAP During Induction
Description: percentage fall in mean arterial pressure from baseline during induction
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: percentage of fall from baseline
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
percentage of fall from baseline | 18.5 (13) | 24 (8)

15. Other Pre Specified Outcome: Total Propofol Used (mg/kg/hr)
Description: total propofol used based on per kg body weight per hour for the whole duration of surgery
Time Frame: 8 hours (approx)
Measure: Mean (Standard Deviation); unit: mg per kg body weight per hour
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
mg per kg body weight per hour | 4.81 (1.98) | 6 (2)

16. Other Pre Specified Outcome: Total Fentanyl Used (µg/kg)
Description: total fentanyl used in the whole duration of surgery on per kg body weight basis
Time Frame: 8 hours(approx)
Measure: Mean (Standard Deviation); unit: microgram per kg body weight
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
microgram per kg body weight | 12.03 (4.51) | 12.5 (4.31)

17. Other Pre Specified Outcome: Total Off CPB Propofol Used (mg/kg/hr
Description: total dosage of propofol used on per kg body weight per hour basis in the period before and after cardiopulmonary bypass period.
Time Frame: 6 hours(approx)
Measure: Mean (Standard Deviation); unit: mg per kg body weight per hour
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
mg per kg body weight per hour | 6.29 (2.48) | 7.82 (2.1)

18. Other Pre Specified Outcome: Number of Times Rate of Propofol Changed Manually
Description: Number of times rate of propofol needed to be changed manually
Time Frame: 8 hours(aprrox)
Measure: Median (Full Range); unit: times per hour
Arm/Group | IAADS Group | Manual Group
Number analyzed (Participants) | 20 | 20
times per hour | 0 [0 to 0] | 18 [8 to 29]

ADVERSE EVENTS:
Arm/Group | IAADS Group | Manual Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
anesthesiologist could get visual impression of his performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No